CLINICAL TRIAL: NCT03040687
Title: Protective Efficacy of Orally Delivered Bovine Serum Immunoglobulin (BSIgG) Specific for the Colonization Factor CS6 Following Challenge With the CS6-expressing Enterotoxigenic E. Coli (ETEC) Strain B7A
Brief Title: Efficacy of B7A BSIgG Against E. Coli Strain B7A Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIR 315 BSIgG
Record Dates: First submitted 2017-01-26; First posted 2017-02-02 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteer
Keywords: ETEC; Escherichia coli; enteritis; challenge; CS6; B7A
MeSH Terms: conditions — Escherichia coli Infections; Enteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anti-CS6 group (Experimental): Anti-CS6 BSIgG and challenge strain CS6-expressing ETEC (B7A)
  Interventions: Biological: Anti CS6 BSIgG product (Lot PD1601105CS); Biological: B7A- CS6-expressing ETEC challenge strain
- Anti-whole cell B7A (Experimental): Anti- whole cell B7A (killed) BSIgG and challenge strain CS6-expressing ETEC (B7A)
  Interventions: Biological: Anti B7A BSIgG product (Lot PD1601132ET); Biological: B7A- CS6-expressing ETEC challenge strain
- control Immunoglobulin group (Experimental): Negative Control (Nonhyperimmune BSIgG placebo) and challenge strain CS6-expressing ETEC (B7A)
  Interventions: Biological: Bovine Immunoglobin Negative Control (Lot PD161071NC); Biological: B7A- CS6-expressing ETEC challenge strain

INTERVENTIONS:
Biological: Anti CS6 BSIgG product (Lot PD1601105CS)
  Arms: Anti-CS6 group
Biological: Anti B7A BSIgG product (Lot PD1601132ET)
  Arms: Anti-whole cell B7A
Biological: Bovine Immunoglobin Negative Control (Lot PD161071NC)
  Arms: control Immunoglobulin group
Biological: B7A- CS6-expressing ETEC challenge strain

SUMMARY:
Enterotoxigenic Escherichia coli (ETEC) is a major cause of diarrhea worldwide. Vaccines and therapeutics are under development to prevent ETEC disease in children and travelers. One approach is to use passive protection (antibodies) to prevent infection. The purpose of this study are to assess the safety of serum-derived bovine immunoglobulins in healthy adult subjects when orally administered and to estimate protective efficacy of those preparations against moderate-severe diarrhea upon challenge with the ETEC strain B7A.

DETAILED DESCRIPTION:
Enterotoxigenic Escherichia coli (ETEC) is one of the most common causes of infectious diarrhea in children in resource limited countries, and is also a frequent cause of traveler's diarrhea in civilian and military travelers to endemic countries. ETEC strains express a variety of colonization factors (CF) that help them attach to the intestinal wall. Each colonization factor has one or more surface antigens (CS). One of the major surface antigens of ETEC is CS6 (Coli surface antigen 6).

Vaccines and treatments to prevent ETEC disease are under development. Some of these target specific enterotoxins or colonization factors. For over 40 years, we have used ETEC human challenge studies to understand the ETEC disease process, immune response, and more recently, to determine whether treatments or vaccines are protective or effective in mitigating disease. B7A is the only CS6 expressing ETEC challenge strain currently used.

A modality that has shown some success in the prevention of diarrhea is passive, oral administration of bovine milk IgG with specific activity against viral, bacterial and parasitic enteropathogens. Passive oral administration of Bovine Serum Immunoglobulins (BSIgG) may protect against ETEC-mediated infectious diarrhea. The hypothesized mechanism of protection stems from the passive administration of bovine anti-tip adhesion or fimbriae antibodies preventing their adherence in the human small intestine (the initial step in pathogenesis), thereby preventing downstream pathogenic processes and symptomatic illness. This study will establish the foundation for evaluating BSIgG products against numerous ETEC CFs.

This study will explore if anti-B7A and anti- CS6 BSIgG provides protection against oral challenge with B7A in healthy adult volunteers. There will be two inpatient admissions of approximately 30 subjects (up to 60 total). They will receive one of three investigational products (IP) three times daily following meals beginning 2 days prior to challenge. Each volunteer will be challenged with CS6 expressing ETEC B7A on Day 0. The investigational product/placebo will be administered for a total of 7 days, or until antibiotic treatment has been administered. The investigators hypothesize that anti-CS6 BSIgG will provide protection against B7A mediated moderate to severe diarrhea upon challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 50 years of age, inclusive.
* General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by principal investigator (PI) or PI in consultation with the research monitor and sponsor.
* Demonstrate comprehension of the protocol procedures and knowledge of ETEC illness by passing a written examination (pass grade ≥ 70%)
* Willing to participate after informed consent obtained.
* Available for all planned follow-up visits.
* Negative serum pregnancy test at screening and negative serum and/or urine pregnancy test on the day of admittance to the inpatient phase for female subjects of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female subjects unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).

Exclusion Criteria:

General health criteria

* Presence of a significant medical condition, (e.g. psychiatric conditions or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease, alcohol or illicit drug abuse/dependency, or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
* Immunosuppressive illness or Immunoglobulin A (IgA) deficiency (serum IgA < 7 mg/dL or below the limit of detection of assay)
* Evidence of confirmed infection with HIV, HBsAg, or Hepatitis C Virus (HCV), with confirmatory assays.
* Use of any investigational product within 30 days preceding the receipt of the investigational products, or planned use during the active study period
* Significant abnormalities in screening lab hematology or serum chemistries, as determined by PI or PI in consultation with the research monitor and sponsor.
* Lactation or breastfeeding.

Research-related exclusions applicable to challenge

* History of microbiologically confirmed ETEC or cholera infection in last 3 years.
* Occupation involving handling of ETEC or Vibrio cholerae currently, or in the past 3 years.
* Travel to countries where ETEC or cholera infection is endemic (most of the developing world) within 3 years prior to dosing.
* Symptoms consistent with Travelers' Diarrhea concurrent with travel to countries where ETEC infection is endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study.
* Vaccination for or ingestion of ETEC, cholera, or E coli heat labile toxin within 3 years prior to dosing.
* Any prior experimental infection with ETEC strain B7A.

Study-specific Exclusion Criteria (potential increased risk or complicating outcome ascertainment)

* Abnormal stool pattern (fewer than 3 per week or more than 3 per day).
* History of diarrhea in the 2 weeks prior to planned inpatient phase.
* Regular use of laxatives, antacids, or other agents to lower stomach acidity (regular defined as at least weekly).
* Use of antibiotics during the 7 days before receipt of any investigational

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R Talaat, MD, Principal Investigator — Johns Hopkins Center for Immunization Research
Locations (1):
- Johns Hopkins Center for Immunization Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Porter CK, Riddle MS, Alcala AN, Sack DA, Harro C, Chakraborty S, Gutierrez RL, Savarino SJ, Darsley M, McKenzie R, DeNearing B, Steinsland H, Tribble DR, Bourgeois AL. An Evidenced-Based Scale of Disease Severity following Human Challenge with Enteroxigenic Escherichia coli. PLoS One. 2016 Mar 3;11(3):e0149358. doi: 10.1371/journal.pone.0149358. eCollection 2016. PMID 26938983
- [Background] McKenzie R, Porter CK, Cantrell JA, Denearing B, O'Dowd A, Grahek SL, Sincock SA, Woods C, Sebeny P, Sack DA, Tribble DR, Bourgeois AL, Savarino SJ. Volunteer challenge with enterotoxigenic Escherichia coli that express intestinal colonization factor fimbriae CS17 and CS19. J Infect Dis. 2011 Jul 1;204(1):60-4. doi: 10.1093/infdis/jir220. PMID 21628659
- [Background] Freedman DJ, Tacket CO, Delehanty A, Maneval DR, Nataro J, Crabb JH. Milk immunoglobulin with specific activity against purified colonization factor antigens can protect against oral challenge with enterotoxigenic Escherichia coli. J Infect Dis. 1998 Mar;177(3):662-7. doi: 10.1086/514227. PMID 9498445

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty healthy adult naive subjects enrolled and received one of the three BSIgG products. Fifty-nine of those subjects were challenged with ETEC strain B7A.
Pre-assignment Details: Study specific screening occurred prior to enrollment. Eighty-two subjects signed study specific consent forms. Nineteen subjects screened failed. Three subjects were randomized but did not receive BSIgG.
Groups:
- Anti-CS6 Group: Anti-CS6 BSIgG and challenge strain CS6-expressing ETEC (B7A)
  Anti CS6 BSIgG product (Lot PD1601105CS)
  B7A- CS6-expressing ETEC challenge strain
- Anti-whole Cell B7A: Anti- whole cell B7A (killed) BSIgG and challenge strain CS6-expressing ETEC (B7A)
  Anti B7A BSIgG product (Lot PD1601132ET)
  B7A- CS6-expressing ETEC challenge strain
- Control Immunoglobulin Group: Negative Control (Nonhyperimmune BSIgG placebo) and challenge strain CS6-expressing ETEC (B7A)
  Bovine Immunoglobin Negative Control (Lot PD161071NC)
  B7A- CS6-expressing ETEC challenge strain
Period: Overall Study
Arm/Group | Anti-CS6 Group | Anti-whole Cell B7A | Control Immunoglobulin Group
Started | 20 | 20 | 20
Completed | 19 | 20 | 20
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-CS6 Group | Anti-whole Cell B7A | Control Immunoglobulin Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.5 [25.0 to 37.5] | 35.0 [31.0 to 43.0] | 35.5 [26.8 to 41.8] | 34 [26.8 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 9 | 22
  Male | 11 | 16 | 11 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 3 | 7
  Not Hispanic or Latino | 17 | 19 | 17 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 18 | 15 | 48
  White | 5 | 2 | 3 | 10
  More than one race | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Safety of Serum Derived Bovine Immunoglobulins (BSIgG)
Description: Number of Participants with adverse events in groups receiving B7A- and CS6- hyperimmune (BSIgG) compared with the group receiving the nonhyperimmune product.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-CS6 Group | Anti-whole Cell B7A | Control Immunoglobulin Group
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Abdominal Distension | 1 | 2 | 0
  Abdominal Pain | 2 | 0 | 1
  Defecation Urgency | 0 | 0 | 1
  Flatulence | 3 | 4 | 2
  Headache | 0 | 2 | 0
  Nausea | 0 | 1 | 0
  None | 14 | 11 | 16

2. Primary Outcome: Efficacy of B7A and CS6- Hyperimmune Bovine Serum Immunoglobin to Protect Against Moderate to Severe Diarrhea After Challenge With the CS6 Expressing ETEC Strain B7A
Description: Comparison of the number and percentage of volunteers in the arms receiving the B7A- and CS6 BSIgG vs the arm receiving the nonhyperimmune BSIgG who develop moderate to severe diarrhea.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-CS6 Group | Anti-whole Cell B7A | Control Immunoglobulin Group
Number analyzed (Participants) | 19 | 20 | 20
Participants | 12 | 7 | 14

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Anti-CS6 Group | Anti-whole Cell B7A | Control Immunoglobulin Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/20 | 17/20 | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-CS6 Group (N=20) | Anti-whole Cell B7A (N=20) | Control Immunoglobulin Group (N=20)
Abdominal Distention (Gastrointestinal disorders) | 2 (2) | 2 (2) | 9 (9)
Abdominal Pain (Gastrointestinal disorders) | 12 (12) | 7 (7) | 12 (12)
Abdominal Pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 5 (5) | 0 (0) | 7 (7)
Apthous ulcer (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthraligia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (Immune system disorders) | 7 (7) | 0 (0) | 5 (10)
Decreased appetite (Gastrointestinal disorders) | 10 (10) | 4 (4) | 10 (10)
Defecation Urgency (Gastrointestinal disorders) | 9 (9) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT03040687/Prot_SAP_000.pdf